CLINICAL TRIAL: NCT06060405
Title: Durvalumab and Oleclumab in Resectable PDAC: A Window of Opportunity Study (DORA Trial)
Brief Title: Durvalumab and Oleclumab in Resectable PDAC
Acronym: DORA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZUHN-013; 22-6031 (Other: University Health Network)
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab and Oleclumab (Experimental): Durvalumab, 1500 mg x 1 dose and oleclumab 3000 mg x 2 doses every 2 weeks prior to surgical resection.
  Interventions: Drug: Durvalumab; Drug: Oleclumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is a monoclonal antibody that blocks the interaction of PD-L1 with PD-1 on immune cells.
  Other Names: IMFINZI
Drug: Oleclumab — Oleclumab is a monoclonal antibody that binds to and inhibits the activity of CD73.
  Other Names: MEDI9447

SUMMARY:
This is a multi-site Canadian, window of opportunity study to evaluate the immune activity of durvalumab and oleclumab in resectable pancreatic ductal adenocarcinoma (PDAC) when given prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Weight ≥ 35 kg
* Have a life expectancy ≥ 12 weeks
* Have histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC).
* Upfront resectable PDAC
* Have adequate organ and marrow function required for the study
* Baseline images taken prior to treatment must undergo central review
* Participants must agree to use study approved methods to prevent pregnancy for study required period

Exclusion Criteria:

* Receipt of any conventional or investigational anticancer therapy within 21 days or palliative radiotherapy within 14 days prior to the scheduled first dose of study treatment
* Prior receipt of any immune-mediated therapy including, but not limited to, other anti CTLA-4, anti-PD-1, anti-PD-L1 including durvalumab antibodies and agents targeting CD73, CD39, or adenosine receptors, excluding therapeutic anticancer vaccines.
* Concurrent enrolment in another therapeutic clinical study. Enrolment in observational studies will be allowed.
* Have a history of Grade 3 or greater thromboembolic events in the prior 3 months or thromboembolic event of any grade with ongoing symptoms.
* Have prior history of myocardial infarction, transient ischemic attack, congestive heart failure ≥ Class 3 based on New York Heart Association Functional Classification or stroke within the past 3 months prior to the scheduled first dose of study treatment.
* Active or prior documented autoimmune disorders within the past 3 years prior to the scheduled first dose of study treatment with the following exceptions

  * Vitiligo or alopecia
  * Hypothyroidism not requiring systemic treatment or stable on hormone replacement
  * Psoriasis not requiring systemic treatment
  * Any chronic skin condition that does not require systemic therapy
* Have known active hepatitis infection. Participants with a past or resolved Hepatitis B (HBV) infection are eligible. Participants positive for Hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection
* Other invasive malignancy within 5 years.
* Known allergy or hypersensitivity to investigational product formulations.
* Active grade 3 or greater edema
* Uncontrolled intercurrent illness
* Current or prior use of immunosuppressive medication within 14 days prior to the scheduled first dose of study treatment with the following exceptions:

  * Intranasal, topical, inhaled corticosteroids or local steroid injections
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reaction
* Receipt of live, attenuated vaccine within 30 days prior to the scheduled first dose of study treatment
* Major surgery within 28 days prior to scheduled first dose of study treatment or still recovering from prior surgery. Local are allowed, without needing to wait for the 28 day recovery period.
* Are pregnant, lactating, or intend to become pregnant during their participation in the study
* Any condition that, in the opinion of the investigator, would interfere with safe administration or evaluation of the investigational products or interpretation of subject safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in CD8+ cell infiltration | Baseline biopsy to surgical resection (35 days)

SECONDARY OUTCOMES:
Percent change in CD3 cell population in tumour tissue | Baseline biopsy to surgical resection (35 days)
Percent change in CD3 cell population in blood | Baseline biopsy to surgical resection (35 days)
Percent change in CD45RA cell population in tumour tissue | Baseline biopsy to surgical resection (35 days)
Percent change in CD45RA cell population in blood | Baseline biopsy to surgical resection (35 days)
Percent change in RO T cell population in tumour tissue | Baseline biopsy to surgical resection (35 days)
Percent change in RO T cell population in blood | Baseline biopsy to surgical resection (35 days)
Percent change in M1 vs M2 macrophage population in tumour tissue | Baseline biopsy to surgical resection (35 days)
Percent change in M1 vs M2 macrophage population in blood | Baseline biopsy to surgical resection (35 days)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Moore, MD, Principal Investigator — Princess Margaret Cancer Centre/University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada